CLINICAL TRIAL: NCT06844084
Title: Biopsychosocial Effects of Gardening Activities on Elderly People in Nursing Homes
Brief Title: Biopsychosocial Effects of Gardening Activities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Asos.Prof., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OrduBAP
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cognition; Anxiety; Depression; Life Satisfaction; Psychological Well Being
Keywords: Elderly; Gardening Activity; Psychological Well Being; Anxiety; Depression; Life Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Depression; Personal Satisfaction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study was planned as a single-blind randomized controlled experimental study. Randomized controlled experimental studies are the research design that is the source of evidence-based information on the applicability of a particular intervention, determines causality and is the basic source for systematic reviews and meta-analyses that are evaluated as first-level evidence. In this project, a randomized controlled study design was chosen to examine the biopsychosocial effects of gardening activities applied to elderly people in nursing homes and to obtain high-level evidence results. Blinding is performed to prevent bias in randomized controlled studies (Akın and Koçoğlu, 2017). In this project, participants and analyzers can be blinded to prevent bias, therefore, the study was planned to be conducted in a single-blind randomized controlled experimental design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the project, gardening activities will be applied to the participants in the experimental group once a week for 60 minutes for 16 weeks (4 months) in a nursing home and greenhouse. In the project, the elderly will be informed about gardening activities in the nursing home. The applications will be carried out in the greenhouse.
  Interventions: Other: Gardening Activity
- Control Group (No Intervention): Participants in the control group will not receive any intervention during the study. They will participate in routine activities in the nursing home (crafts such as philography, relief, knitting, and folk dances and bocce games in the atelier). After the final tests are administered in the study, participants in the control group will be engaged in gardening activities for 60 minutes once a week for 4 weeks (1 month) (this period was determined by taking the project duration into account).

INTERVENTIONS:
Other: Gardening Activity — In the project, gardening activities will be applied to the participants in the experimental group in the nursing home and greenhouse for 16 weeks (4 months), once a week for 60 minutes. During the implementation phase of horticulture activities, information meetings will be held in the meeting room of the nursing home in one group. In addition, 20 minutes break will be given during the activity in terms of the tolerance of the elderly to gardening activities.
  Arms: Experimental Group

SUMMARY:
Due to the increasing number of elderly population worldwide, elderly care is becoming increasingly important and the number of elderly in institutional care is increasing. In this context, the implementation of easily applicable, cost-effective and accessible physical activity programmes for the elderly in nursing homes is important for the physical, mental and social health of the elderly. Gardening activities are a non-pharmacological intervention that has recently increased in popularity in the elderly and can be easily applied. It is known that gardening activities in the elderly affect some biochemical parameters along with mental health effects and reduce stress, especially by reducing cortisol levels. By providing physical mobility in the elderly with gardening activities, there may be an increase in irisin level and BDNF level, which is an indicator of improvement in cognitive functions, and a decrease in cortisol level, which is an indicator of stress. With the project, the effects of gardening activities on the elderly will be examined comprehensively in a biopsychosocial manner. In this project, the effects of gardening activities on anxiety, depression, life satisfaction, psychological well-being and biochemical parameters will be examined in the elderly living in a nursing home. In the project, gardening activities will be applied to the elderly in the experimental group once a week for 60 minutes for 16 weeks (4 months). With the project, it is aimed to strengthen the elderly biopsychosocially by making them do gardening activities.

DETAILED DESCRIPTION:
Improvement of living conditions, development of health services and technology lead to prolonged life expectancy and accordingly, the number of elderly population is gradually increasing. For this reason, elderly care is becoming increasingly important and the number of elderly in institutional care is increasing. The elderly in nursing homes may experience many physical, mental and social problems. The elderly in nursing homes may experience problems such as decreased self-esteem, increased dependency in daily living activities, chronic diseases, fear of death, lack of social support, cognitive deficiencies, anxiety due to environmental and lifestyle changes, depression and lack of life satisfaction. In this context, the implementation of easily applicable, cost-effective and accessible physical activity programmes for the elderly in nursing homes is important for the physical, mental and social health of the elderly. Gardening activities are a non-pharmacological intervention that has recently increased in popularity in the elderly and can be easily applied. Gardening activities positively affect the sense of commitment and success, self-expression, social interaction, sense of responsibility, self-esteem, cognitive skills and creativity in the elderly. It is known that gardening activities in the elderly affect some biochemical parameters along with mental health effects and reduce stress, especially by reducing cortisol levels. By providing physical mobility in the elderly with gardening activities, there may be an increase in irisin level and BDNF level, which is an indicator of improvement in cognitive functions, and a decrease in cortisol level, which is an indicator of stress. In the literature, it is seen that studies examining the effects of gardening activities on the health of the elderly have been carried out, but the studies on this subject in our country are very limited. With the project, for the first time in our country, the effects of gardening activities on the elderly will be examined comprehensively in a biopsychosocial manner. In this project, the effects of gardening activities on anxiety, depression, life satisfaction, psychological well-being and biochemical parameters will be examined in the elderly living in a nursing home. In the project, gardening activities will be applied to the elderly in the experimental group once a week for 60 minutes for 16 weeks (4 months). With the project, it is aimed to strengthen the elderly biopsychosocially by making them do gardening activities.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people who have been living in a nursing home for at least 6 months,
* Elderly people with a mini mental test score of 24 and above,
* Elderly people who do not have vision or hearing loss that may prevent gardening activities,
* Elderly people who are open to communication and cooperation and who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Elderly people with physical (such as stroke, Parkinson's) and psychiatric diseases (such as mental retardation) that may prevent gardening activities,
* Elderly people with chronic diseases in the exacerbation process (heart failure, chronic renal failure, etc.) will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Geriatric Anxiety Inverntory | At the beginning of the study and end of 16 weeks treatment
  The scale developed by Pachana et al. (2007) was adapted to Turkish by Pamir Akın (2010). The Geriatric Anxiety Inventory aims to measure anxiety symptoms in the elderly in a dimensional manner. The cut-off point of the scale for generalized anxiety disorder was determined as 10/11. Accordingly, the scale was organized as "anxiety symptoms and generalized anxiety disorder > 10; only anxiety symptoms < 10". There are no reverse-coded items in the scale, which consists of 20 items and is scored on two dimensions as "agree" and "disagree". Accordingly, 1 point is given for the "agree" option and 0 points for the "disagree" option. Therefore, the scores obtained from the scale can vary between 0 and 20. Cronbach's α for the normal elderly sample was found to be 0.91, and Cronbach's α for the psychogeriatric sample was found to be 0.93.
Geriatric Depression Scale | At the beginning of the study and end of 16 weeks treatment
  The scale developed by Yesavage et al. (1993) is based on self-reporting. The short form of the GDS consisting of 15 questions will be used in this study. The Turkish validity and reliability study of the scale was conducted by Ertan et al. (1997). 5 questions (1, 5, 7, 11 and 13) in the scale were designed positively, the others were designed negatively. In the evaluation of the scale, "no" answers to positive questions and "yes" answers to negative questions were matched with 1 point. The scores that can be obtained from the scale are between 0-15. A score above five is considered depression. The Cronbach alpha value of the scale is 0.92.
Life Satisfaction in the Elderly Scale | At the beginning of the study and end of 16 weeks treatment
  The scale was developed by Altay and Çalmaz (2022) and consists of a total of 14 items and 3 sub-dimensions. The scale was prepared as a Likert-type, five-point scale (1= Strongly disagree, 2= Disagree, 3= Neither agree nor disagree, 4= Agree, 5= Strongly agree). The score that can be obtained from ELS varies between 14 and 70. A high score indicates that the individual has high life satisfaction. ELS contains a three-factor structure. Self-acceptance (Factor 1) of the sub-dimensions of the scale includes items 5, 6, 8, 9, 16, 21, 25, 27, 28, Motivation (Factor 2) includes items 11 and 13, and Peace (Factor 3) includes items 10, 12, and 14. Sub-dimension scores are calculated by adding the scores of the items in each sub-dimension and dividing them by the number of items. Each sub-dimension is scored between '1' and '5'. The self-acceptance sub-dimension score range is minimum - maximum 9-45, the motivation sub-dimension score range is minimum - m
Psychological Well-Being Scale for Older People | At the beginning of the study and end of 16 weeks treatment
  It was developed by Gümüş Demir (2022) to measure happiness and well-being in elderly individuals, and has a 15-item and single-factor structure. Items 8 and 13 are reverse coded. The single-factor structure of the scale was tested in a different sample group with the CFA method and the result that the structure was confirmed was obtained. The scale was found to be a valid and reliable measurement tool for measuring psychological well-being in the elderly. The Cronbach alpha internal consistency coefficient of the scale was found to be 0.89.

IPD SHARING:
Plan to Share IPD: No